CLINICAL TRIAL: NCT01603862
Title: Piloting a Complex Intervention Involving Physical Exercise, Cognitive Training and Socialising to Delay the Onset of Dementia in Mild Cognitive Impairment
Brief Title: ThinkingFit: Combined Physical, Cognitive and Social Treatment in Mild Cognitive Impairment (MCI)
Acronym: ThinkingFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Thomas Dannhauser (Other Government)
Collaborators: University College, London (Other)
Responsible Party: Sponsor-Investigator, Dr Thomas Dannhauser, Consultant Psychiatrist and Honorary Senior Lecturer in Psychiatry, North Essex Partnership NHS Foundation Trust
Organization: North Essex Partnership NHS Foundation Trust (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThinkingFit 1
Record Dates: First submitted 2012-05-17; First posted 2012-05-23 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ThinkingFit (Experimental)
  Interventions: Procedure: ThinkingFit programme

INTERVENTIONS:
Procedure: ThinkingFit programme — Combined physical, cognitive and social stimulation activties.

SUMMARY:
Dementia is serious problem and around 700 000 people are affected in the UK alone. Currently there is no cure however early diagnosis and effective treatment offers hope for reducing the impact. Dementia sufferers require care due to physical disability, cognitive deficits, social isolation and emotional symptoms (depression). Delaying the onset of dementia will improve quality of life for patients and reduce the cost of residential care (£42 000 per person per year).

People with mild cognitive impairment (MCI) are at high risk of developing dementia. They have impaired cognitive abilities, such as memory, but still manage their everyday activities. Studies show that 8 out of 10 people with MCI will have developed dementia 6 years after diagnosis.

Regular physical activities and performing a variety of cognitive activities reduce the risk of dementia and improves abilities and quality of life in healthy people. Therefore a combination of these activities may reduce the risk of developing dementia in MCI. The investigators want to see if they can develop a program which combines these activities in a fun and social way that gets people active and keeps them active. The aims are to improve fitness, cognition and quality of life. The investigators plan to use computers and the internet to help with the activities and to make them available to people who are isolated. Physical activity will involve walking from home, cognitive activities will be computer based games and puzzles and socialising will involve regular varied group-based activities. Participants (128) will be recruited from the UCL Derwent Memory Clinic and will complete a 26 week program. They will then be followed up yearly to monitor their progress. The main outcome of the study is engagement in the activities. The investigators will also measure fitness, cognition, quality of life and conversion to dementia.

ELIGIBILITY:
Inclusion criteria for patients with MCI

1. Patients fulfilling criteria for AMCI [Petersen et al. 2001b]:

   i. Memory impairment for age and education ii. No impairment in other cognitive domains iii. Normal social activities iv. Patient is not demented
2. For the other subtypes of MCI, cognitive impairment in one or more nonmemory domain
3. Sedentary lifestyle with no regular participation in physical exercise defined as two or three times a week for at least 20 minutes duration, or participation in active sport more than once a week, in the previous six months.
4. Willing and able to give informed consent.
5. Availability and access to safe exercise environments, such as paths or roads with sidewalks for walking or cycling.
6. At low risk from serious adverse effects from increased physical activity as indicated by performance on the revised Physical activity readiness questionnaire (PARQ).

Exclusion Criteria:

Exclusion criteria for patients with MCI

1. Type 1 (insulin dependent) diabetes mellitus.
2. Blood pressure of 160/100 mmHg or more.
3. Body weight more than 140% of ideal body weight.
4. Musculoskeletal or other medical problems preventing safe participation in regular moderate intensity exercise (65-77% of predicted maximum heart rate). This will include a resting tachycardia (heart rate above 100 bpm) and history of myocardial infarction or unstable angina within the last month.

Participants with modifiable exclusion criteria will be reconsidered after successful management. Patients will be referred for medical treatment prior to commencing exercise if indicated by the PARQ and the intervention will be guided by the PARmedX.

Participants taking medications affecting heart rate will need to be on a stable dosing regime for 3 months prior to commencing in order to control for potential spurious results on fitness measures caused by these treatments.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Activity Compliance | Compliance with programmed activities will be assessed at the end of participation which is expected to be at 24 weeks
  Number of participants to have completed 50% or more of the programmed activity sessions during the intervention period.

SECONDARY OUTCOMES:
Cardiovascular fitness measure | This will be measured at the start, after the control period (12 weeks) and after completion of the activity interventions at around 24 weeks.
  Cardiovascular fitness will be measured with a modified Siconolfi Step Test.
Cognitive measures | This will be measured at the start, after the control period (12 weeks) and after completion of the activity interventions at around 24 weeks.
  Participants will complete the following cognitive measures:
  * Visual and auditory divided attention task
  * Verbal episodic encoding and recognition task
  * Halstead Trail Making test (TMT)
  * Verbal fluency
  * Working memory tests: digit span forwards/ backwards
Measures of quality of life and everyday activities | This will be measured at the start, after the control period (12 weeks) and after completion of the activity interventions at around 24 weeks.
  Quality of life will be measured on the World Health Organization Quality of Life (WHOQOL) - BREF and change in every day activities on the Alzheimer's Disease Cooperative Study MCI Activities of Daily Living Scale (ADCS-MCI-ADL)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Cleverley, Principal Investigator — North Essex Partnership Foundation NHS Trust; Thomas M Dannhauser, PhD, Study Director — University College London, North Essex Partnership NHS Foundation Trust
Locations (1):
- North Essex Partnership Foundation NHS Trust, Harlow, Essex, United Kingdom

REFERENCES:
- [Derived] Dannhauser TM, Cleverley M, Whitfield TJ, Fletcher BC, Stevens T, Walker Z. A complex multimodal activity intervention to reduce the risk of dementia in mild cognitive impairment--ThinkingFit: pilot and feasibility study for a randomized controlled trial. BMC Psychiatry. 2014 May 5;14:129. doi: 10.1186/1471-244X-14-129. PMID 24886353